CLINICAL TRIAL: NCT00902798
Title: Cognitive Enhancement Therapy for Adult Autism Spectrum Disorder
Acronym: Perspectives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Autism Speaks (Other); United States Department of Defense (U.S. Federal Agency); Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Shaun M. Eack, Professor of Social Work and Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH085851; R33MH085851 (NIH); R21MH085851 (NIH); AR100344 (Other Grant/Funding Number: Department of Defense); 05381 (Other Grant/Funding Number: Autism Speaks); 2008NF-Autism (Other Grant/Funding Number: Pennsylvania Department of Health); ARI2014 (Other Grant/Funding Number: Autism Research Institute)
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Autistic Disorder; Autism Spectrum Disorder; Asperger's Syndrome; Pervasive Developmental Disorder
Keywords: Autism; Autism Spectrum Disorders; Asperger's Syndrome; Pervasive Developmental Disorder; Cognition; Social Cognition; Psychosocial Treatment; Cognitive Enhancement Therapy; Enriched Supportive Therapy; Therapy; Psychotherapy
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Asperger Syndrome; Child Development Disorders, Pervasive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Enhancement Therapy (Experimental): This research treatment aims to help with problems in thinking, planning, and socialization. Participants begin with cognitive training using computer software programs. They also participate in a small social-cognitive group to learn about their condition and how to act wisely in social situations by developing the abilities needed to understand another person's perspective, evaluate social contexts, and be foresightful.
  Time commitment: about 3½ hours per week; Location: Pittsburgh, PA only
  Interventions: Behavioral: Cognitive Enhancement Therapy
- Enriched Supportive Therapy (Active Comparator): This research treatment uses individual supportive therapy to help adults learn about autism spectrum disorder, manage their emotions and stress, improve their social skills, and cope with everyday problems. Participants will learn about the impact of stress on their lives, and how to identify their own early cues of distress and apply effective coping strategies.
  Time commitment: about 1 hour per week; Location: Pittsburgh, PA only
  Interventions: Behavioral: Enriched Supportive Therapy

INTERVENTIONS:
Behavioral: Cognitive Enhancement Therapy — An 18-month comprehensive, small group approach for the remediation of cognitive deficits in neurodevelopmental disorders consisting of individual sessions and 45 group training sessions in social cognition that are integrated with approximately 60 hours of computer assisted training in attention, memory, and problem solving skills.
  Arms: Cognitive Enhancement Therapy
Behavioral: Enriched Supportive Therapy — An 18-month intervention that uses individual supportive therapy to help adults learn about autism spectrum disorder, manage their emotions and stress, improve their social skills, and cope with everyday problems. Participants will learn about the impact of stress on their lives, and how to identify their own early cues of distress and apply effective coping strategies.
  Arms: Enriched Supportive Therapy

SUMMARY:
This study will investigate and contrast the effects of two psychological treatments for adults with autism spectrum disorder. Cognitive Enhancement Therapy (CET) is a cognitive remediation intervention that aims to help adults with problems in thinking, planning, and socialization. Enriched Supportive Therapy (EST) is an individual supportive therapy that aims to help adults learn about their condition, manage their emotions and stress, improve their social skills, and cope with everyday problems.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is characterized by marked impairments in social and non-social cognitive ability that persist well into adulthood and contribute to significant functional disability. The treatment of ASD has focused almost exclusively on children, and few empirically supported interventions are available to address the core cognitive and functional challenges individuals with ASD face as they transition to adulthood. This study will investigate and contrast the effects of two psychological treatments for adults with autism spectrum disorder. Cognitive Enhancement Therapy (CET) is a cognitive remediation intervention that aims to help adults with problems in thinking, planning, and socialization. Enriched Supportive Therapy (EST) is an individual supportive therapy that aims to help adults learn about their condition, manage their emotions and stress, improve their social skills, and cope with everyday problems.

Participation in this study will last 30 months. Potential participants must be able to attend weekly treatment sessions in Pittsburgh, PA.

The study design is a 30-month (2.5 years) randomized-controlled trial, where eligible participants will be randomized to the CET or EST study treatments. Participants will be treated with the study interventions for 18 months, and then followed for 12 additional months to assess the lasting impact of the study interventions. All participants will complete cognitive, clinical, and neuroimaging (magnetic resonance imaging) assessments prior to starting the study treatments and then at specified intervals thereafter to evaluate the impact of the study treatments on cognition, adaptive function, and the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-45 years
* Diagnosis of autism, Asperger's syndrome, or pervasive developmental disorder not otherwise specified (NOS) verified by the autism diagnostic observation schedule (ADOS) or autism diagnostic interview-revised (ADI-R)
* Presence of significant social and cognitive disability, based on the Cognitive Style and Social Cognition Eligibility Interview (Hogarty et al., 2004)
* Intelligence quotient (IQ) greater than 80
* Ability to read and speak fluent English
* Availability of a family member or close friend allowed to provide information on the participant
* Ability to attend weekly treatment sessions in Pittsburgh, PA

Exclusion Criteria:

* Organic brain syndrome
* IQ < 80
* English language skills below a sixth grade level
* Persistent suicidal or homicidal behavior
* History of substance abuse or dependence within the past 3 months
* Comorbid attention deficit hyperactivity disorder (ADHD)
* Comorbid personality disorder
* History of disruptive or violent behavior
* Any magnetic resonance imaging contraindications

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Neurocognition | Pre-treatment, 9, 18, and 30 months
  Composite measure of neuropsychological tests designed to assess neurocognitive function
Social cognition | Pre-treatment, 9, 18, and 30 months
  Composite measure of performance-based and interview tests designed to assess social-cognitive function

SECONDARY OUTCOMES:
Functional outcome | Pre-treatment, 9, 18, and 30 months
  Functional Assessment Battery (Social, Role, Vocational)

CONTACTS AND LOCATIONS:
Overall Officials: Shaun M. Eack, PhD, Principal Investigator — University of Pittsburgh; Nancy J. Minshew, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the National Database for Autism Research

REFERENCES:
- [Background] Hogarty GE, Flesher S, Ulrich R, Carter M, Greenwald D, Pogue-Geile M, Kechavan M, Cooley S, DiBarry AL, Garrett A, Parepally H, Zoretich R. Cognitive enhancement therapy for schizophrenia: effects of a 2-year randomized trial on cognition and behavior. Arch Gen Psychiatry. 2004 Sep;61(9):866-76. doi: 10.1001/archpsyc.61.9.866. PMID 15351765
- [Background] Hogarty GE, Greenwald DP, Eack SM. Durability and mechanism of effects of cognitive enhancement therapy. Psychiatr Serv. 2006 Dec;57(12):1751-7. doi: 10.1176/ps.2006.57.12.1751. PMID 17158490
- [Background] Eack SM, Hogarty GE, Greenwald DP, Hogarty SS, Keshavan MS. Cognitive enhancement therapy improves emotional intelligence in early course schizophrenia: preliminary effects. Schizophr Res. 2007 Jan;89(1-3):308-11. doi: 10.1016/j.schres.2006.08.018. Epub 2006 Oct 19. PMID 17055227
- [Derived] Eack SM, Hogarty SS, Greenwald DP, Litschge MY, Porton SA, Mazefsky CA, Minshew NJ. Cognitive enhancement therapy for adult autism spectrum disorder: Results of an 18-month randomized clinical trial. Autism Res. 2018 Mar;11(3):519-530. doi: 10.1002/aur.1913. Epub 2017 Dec 29. PMID 29286586